CLINICAL TRIAL: NCT06792630
Title: A Study of the Effect of Laughter Therapy on the Mental Health and Quality of Survival of Hematopoietic Stem Cell Transplant Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: QTJC2024057
Record Dates: First submitted 2024-12-27; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Hematologic Malignancy; Hematopoietic Stem Cell Transplant
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In addition, patients in the intervention group were given laughter therapy intervention from the 1st day of HSCT, with the mnemonic "hihihi (pinyin spelling), hahahaha, eggplant eggplant eggplant, qixi qixi qixi qixi, hahahahahahahahaha," 30 times of the mnemonic as a training session, once a day, from the beginning of the transplantation transfusion +1d to the end of the transplantation transfusion +1d, and then to the end of the transplantation. Patients were discharged from the warehouse, and after discharge, patients were centralized on-line laughter therapy intervention, 1 time/week, repeating 30 times of mnemonics, until 1 year after transplantation.
  Interventions: Behavioral: laughter therapy intervention
- Control group (No Intervention): atients in the intervention group and the control group were given standard therapeutic measures as well as routine care during hospitalization and after discharge in accordance with the recommendations of the appropriate treatment guidelines. The control group used routine nursing education and continuity of care after discharge.

INTERVENTIONS:
Behavioral: laughter therapy intervention — In addition, patients in the intervention group were given laughter therapy intervention from the 1st day of HSCT, with the mnemonic "hihihi (pinyin spelling), hahahaha, eggplant eggplant eggplant, qixi qixi qixi qixi, hahahahahahahahaha," 30 times of the mnemonic as a training session, once a day, from the beginning of the transplantation transfusion +1d to the end of the transplantation transfusion +1d, and then to the end of the transplantation. Patients were discharged from the warehouse, and after discharge, patients were centralized on-line laughter therapy intervention, 1 time/week, repeating 30 times of mnemonics, until 1 year after transplantation.
  Arms: Intervention group

SUMMARY:
主要研究目的：

1)探讨笑疗法在造血干细胞移植患者移植心理健康及生存质量中的效果。 次要研究目的：

1. 了解造血干细胞移植患者移植后3个月、6个月、1年内的心理健康变化和生存质量水平；
2. 探讨笑疗法在造血干细胞移植患者预后等结局指标中的应用效果。

DETAILED DESCRIPTION:
本研究将采用单中心、前瞻性的平行随机对照试验对2024年12月1日至2025年12月1日期间首次接受造血干细胞移植的患者进行招募。对照组实施常规护理措施和出院的常规延续护理措施，干预组从移植+1天开始进行笑治疗，住院期间为移植后+1天至出仓，按照笑的口令"hihihi（拼音拼读），哈哈哈，茄子茄子茄子，七喜七喜七喜，哈哈哈哈哈哈"，30遍口令为1次训练，1天进行1次。出仓及出院后，干预组患者集中线上笑疗法干预，1次/周，重复30遍口令，至移植后1年。分别于移植后3个月、6个月、1年对两组患者在预后、疲劳、焦虑及抑郁、幸福感以及创伤后成长、生存质量及结局指标上进行组间比较，明确笑疗法在造血干细胞移植患者心理健康及生存质量中的效果。

ELIGIBILITY:
Inclusion Criteria:

Patients with a pathologically confirmed diagnosis of hematologic malignancy; Patients undergoing their first hematopoietic stem cell transplant; Age ≥ 16 years; Those who have some reading and writing ability; Those who can cooperate in completing the questionnaires and assessments; Informed consent and voluntary participation in the study.

Exclusion Criteria:

Those with severe mental illness or personality disorders; Those who cannot operate a smartphone independently; Those with severe visual and hearing impairments; Those who are critically ill and cannot receive the intervention.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 months, 6 months, and 1 year
  time between the start of randomization and death from any cause
Progression-free survival | 3 months, 6 months, and 1 year
  time between the start of randomization and progression of the tumor in any respect or death from any cause
Time to treatment failure | 3 months, 6 months, and 1 year
  time from start of randomization to withdrawal from the trial, withdrawal may be due to patient refusal, disease progression, death, adverse events